CLINICAL TRIAL: NCT07259018
Title: A Single-arm, Open Label, Single-center Early Feasibility Study of the LuSeed Aneurysm Embolization System in Individuals With Unruptured Intracranial Aneurysms.
Brief Title: LUMENS-1 Canada Early Feasibility Study Clinical Investigation Plan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LuSeed Vascular LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PRT-0000357
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Aneurysm Cerebral; Bifurcation; Unruptured Intracranial Aneurysm; Saccular Aneurysm; Brain Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LuSeed Aneurysm Embolization System (Experimental)
  Interventions: Device: LuSeed Aneurysm Embolization System

INTERVENTIONS:
Device: LuSeed Aneurysm Embolization System — LuSeed Aneurysm Embolization System EFS Canada

SUMMARY:
The primary objective of this clinical investigation is to evaluate the early safety and feasibility of the LuSeed Aneurysm Embolization System for treating unruptured intracranial aneurysms (IA). This is a single-arm, open-label, single-center, interventional study, screening patients approved for treatment of unruptured IAs based on national or international guidelines. Up to 10 eligible subjects meeting inclusion and exclusion criteria and providing consent will be enrolled in a Canadian site.

DETAILED DESCRIPTION:
LuSeed Vascular will sponsor the study and the study will assess early safety and feasibility of the LuSeed Aneurysm Embolization System for the treatment of unruptured intracranial aneurysms (IA).

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated for treatment of unruptured intracranial aneurysms (IA) according to AHA / ASA Guidelines.
2. Age 18-80 years at screening
3. Patients who are suitable for non-emergency endovascular embolization of saccular IAs
4. The IA must have had the following characteristics:

   * IA located in bifurcation in the anterior or posterior circulation
   * IA dimensions appropriate for treatment with LuSeed- Vascular Embolization Device per implant size selection guidelines as outlined in the Instructions for

   Use (IFU) and as follows:
   * IA Width: 2.5-5.5[mm]
   * IA Neck: 2.0-5.0[mm]
   * IA Height: min 4.0 [mm]- device short configuration, min 5.0 [mm]-device long configuration • The AI must meet the definition of a "wide-neck" aneurysm.
5. Patient is willing and able to participate in the study for the duration of the study follow-up and can comply with study requirements
6. Patient able to give their informed consent can be included in this study.

Exclusion Criteria:

1. Ruptured intracranial aneurysm
2. Patient anatomy or physiology considered unsuitable for endovascular treatment as determined by imaging Core Lab
3. Contraindication for arterial access
4. Intracranial aneurysm neck diameter less than 2mm or greater than 5 mm
5. Intracranial aneurysm sac diameter less than 2.5mm or greater than 5.5mm
6. Intracranial aneurysm minimum height less than 4.0 mm
7. Target Intracranial aneurysm contains other devices/implants (e.g., coils)
8. Stenosis of the target IA's parent vessel >50%
9. Known allergy to platinum, nickel, or titanium
10. Known allergy to contrast agents
11. Absolute contraindication to anticoagulation or antiplatelet therapy
12. Anticoagulation medications such as warfarin that cannot be discontinued
13. Pregnant, breastfeeding or planning pregnancy within next 12 months
14. Acute or chronic renal failure (stage III or IV by VARC-3 criteria)
15. Cerebral embolism, stroke, or TIA in past 6 months
16. Myocardial infarction in the past 6 months
17. Any other medical issue within the brain that would preclude device implantation (such as brain surgery, radiation in the target area of intervention from an external beam source, acute traumatic craniocerebral injury, etc.)
18. Patient had any circulatory, neurovascular, cardiovascular, or neurologic conditions that resulted in unstable neurological symptoms at screening.
19. Patient had physical, neurologic or psychiatric conditions which precluded his/her ability to comply with all aspects of the screening, evaluation, treatment, and the postprocedure follow-up schedule.
20. Other medical conditions that cause an inability to comply with study requirements and/or that could increase the risk of neurovascular procedures (e.g., extreme frailty, liver failure, cancer, heart failure, chronic obstructive pulmonary disease, immunosuppression, neural disease, and hematologic disorders etc.)
21. Patient had a life expectancy of less than 12 months.
22. Current participation in another study with investigational devices or drugs that would confound the effect of the study outcomes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 30 Days Post Study Procedure
  Death of any non-accidental cause, Procedure or Device Related Death or Any Major Disabling Stroke *An independent Medical Monitor (IMM) will adjudicate all data used for safety endpoint analyses
Primary Feasibility Endpoint | Day 0
  Technical Success as defined by: a. Success in accessing target intracranial aneurysm (IA) with the LuSeed Aneurysm Embolization System b. Successful visual confirmation of the LuSeed Aneurysm Embolization System Successful deployment and detachment of the LuSeed Aneurysm Embolization System

SECONDARY OUTCOMES:
Secondary Safety Endpoints | 12 months
  Percentage of participants with death of non-accidental cause or device related death, or major disabling stroke at 6 months and 12 months.
Secondary Safety Endpoints | 12 months
  Percentage of participants presenting each component of the safety composite within first 30 days after treatment, 6 months and 12 months
Secondary Safety Endpoints | 12 months
  Percentage of participants with serious adverse events within the first 30 days after treatment, 6 months and 12 months.
Secondary Effectiveness Endpoints | 6-months and 12-months after treatment
  Proportion of subjects with Complete Aneurysm Occlusion immediate post procedure.
Secondary Effectiveness Endpoints | Day-30, 6-months and 12-months
  Change in mRS between baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital - Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Molyneux AJ, Kerr RS, Yu LM, Clarke M, Sneade M, Yarnold JA, Sandercock P; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group. International subarachnoid aneurysm trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomised comparison of effects on survival, dependency, seizures, rebleeding, subgroups, and aneurysm occlusion. Lancet. 2005 Sep 3-9;366(9488):809-17. doi: 10.1016/S0140-6736(05)67214-5. PMID 16139655
- [Background] Brinjikji W, Cloft HJ, Kallmes DF. Difficult aneurysms for endovascular treatment: overwide or undertall? AJNR Am J Neuroradiol. 2009 Sep;30(8):1513-7. doi: 10.3174/ajnr.A1633. Epub 2009 May 20. PMID 19461057
- [Background] Keedy A. An overview of intracranial aneurysms. Mcgill J Med. 2006 Jul;9(2):141-6. PMID 18523626
- [Background] Faluk M, Das JM, De Jesus O. Saccular Aneurysm. 2024 Mar 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557867/ PMID 32491790
- [Background] Bhaskaran G. INTERNATIONAL JOURNAL OF CURRENT MEDICAL AND PHARMACEUTICAL RESEARCH BRAIN (CEREBRAL) ANEURYSM. November 2018;4:3844-8. https://doi.org/10.24327/23956429.ijcmpr20180569.